CLINICAL TRIAL: NCT00275067
Title: A Phase I/II Trial of Arsenic Trioxide and Temozolomide in Combination With Radiation Therapy for Patients With Malignant Gliomas
Brief Title: Arsenic Trioxide, Temozolomide, and Radiation Therapy in Treating Patients With Malignant Glioma That Has Been Removed By Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Cephalon (Industry); CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04C1; NU 04C1 (Other: Northwestern University); CDR0000456504 (Registry Identifier: PDQ); STU00007792 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult gliosarcoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult glioblastoma; adult giant cell glioblastoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Gliosarcoma; Oligodendroglioma; Glioma; Glioblastoma; Brain Neoplasms | interventions — Arsenic Trioxide; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation + temozolomide and arsenic trioxide (Experimental): Radiation therapy followed by the combination of temozolomide and arsenic trioxide at the maximum tolerated dose determined in phase 1
  Interventions: Drug: arsenic trioxide; Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: arsenic trioxide — Arsenic trioxide administered intravenously at a dose of 0.20mg/kg Daily x 5 week then twice per week
  Other Names: ATO; TRISENOX
Drug: temozolomide — Temozolomide administered orally once per day 1 hour prior to radiation therapy at a dose of 75 mg/m2 x 42 days; at a dose of 200mg/m2 for 5 days every cycle (1 cycle = 28 days) after radiation therapy
  Other Names: TMZ; Temodar
Radiation: radiation therapy — All patients will receive 5940-6120 cGy of radiation therapy as 28-33 treatments/fractions (180-200 cGy/treatment) depending on whether they receive standard 3-D conformal radiation therapy or intensity modulated radiation therapy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving arsenic trioxide and temozolomide together with radiation therapy after surgery may kill any remaining tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of arsenic trioxide and temozolomide when given together with radiation therapy and to see how well they work in treating patients with malignant glioma that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of arsenic trioxide and temozolomide when combined with radiotherapy in patients with resected supratentorial malignant glioma. (Phase I)
* Determine the toxicity of this regimen in these patients. (Phase I)

Secondary

* Determine the 6- and 12-month progression-free survival of patients treated with this regimen once an MTD is reached. (Phase II)
* Determine the radiographic response for patients treated with the above regimen. (Phase II)
* Determine the safety of this regimen in these patients. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of arsenic trioxide and temozolomide followed by a phase II study.

* Phase I: Patients undergo radiotherapy once daily 5 days a week and receive oral temozolomide once daily for approximately 6½ weeks. Patients also receive arsenic trioxide IV over 1-4 hours once daily, 5 days a week in week 1 and then twice a week in weeks 2-7. Beginning within 3-5 weeks after completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 1 year in the absence of disease progression and unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of arsenic trioxide and temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients undergo radiotherapy and receive arsenic trioxide and temozolomide as in phase I at the MTD. Patients then receive temozolomide as in phase I for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 12-18 patients will be accrued for the phase I portion of this study. A total of 25 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial malignant glioma of 1 of the following types:

  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed gliomas
  * Anaplastic gliomas not otherwise specified
* Has undergone surgical resection of tumor

  * Patients with biopsy only are eligible
  * Evaluable or measurable disease following resection of recurrent tumor is not mandated for entry into the study
* No brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 3 months
* WBC > 3,000/mm^3
* Absolute neutrophil count > 2,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 10 g/dL (eligibility level for hemoglobin may be reached by transfusion)
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 2 mg/dL
* Transaminases ≤ 2 times the upper limit of normal
* Serum potassium* > 4.0 mEq/dL
* Serum magnesium* > 1.8 mg/dL NOTE: *If these serum electrolytes are below the specified limits on the baseline laboratory tests, supplemental electrolytes should be administered to bring the serum concentrations to these levels before administering arsenic trioxide
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No second-degree heart block
* QT interval ≤ 460 msec
* No other malignancy within the past 3 years except curatively treated carcinoma in situ or basal cell carcinoma of the skin
* Patients who cannot undergo MRI are not eligible for this study
* No other serious concurrent infection or other medical illness that would jeopardize the ability of the patient to receive the therapy in this protocol with reasonable safety

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Patients must have recovered from the effects of surgery prior to the start of treatment (10-14 days minimum) and be maintained on a stable corticosteroid regimen for 5 days
* Concurrent glucocorticoid therapy allowed at the smallest effective dose
* Patients must be on non-enzyme-inducing anti-convulsants to minimize any drug reaction
* No prior radiation therapy, chemotherapy, immunotherapy, therapy with biologic agents (including immunotoxins, immunoconjugates, antisense agents, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphokine-activated killer cells, or gene therapy), or hormonal therapy for their brain tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-05; Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of arsenic trioxide and temozolomide in combination with radiotherapy | Toxicity evaluated prior to each treatment cycle
  Escalating doses of study drug until dose limiting toxicities are observed.
Collect data on the toxicity of arsenic and temozolomide during radiation therapy | Toxicity evaluated prior to each treatment cycle
  Toxicity of this drug combination during radiation therapy will be assessed.
Assess serum biomarkers and correlate with tumor tissue | At baseline, during radiation therapy, and prior to each cycle of chemotherapy
  Blood will be drawn at baseline, during radiation therapy, and prior to each cycle of chemotherapy to assess serum biomarkers and correlate with tumor tissue.

SECONDARY OUTCOMES:
Determine progression free survival at 6 and 12 months | At 6 and 12 months after beginning chemotherapy
  Patients will undergo an MRI and neurological evaluation every 6 months while on chemotherapy.
Determine time to disease progression | At 6 and 12 months after beginning chemotherapy
  Disease status will be assessed by MRI and neurological examination every 6 months until disease progression.
To determine overall survival | Every 6 months while on treatment
  Survival status will be evaluated every 6 months while on treatment.
To determine radiographic response to study regimen | Every 6 months while on treatment
  Radiographic response will be assessed by MRI every 6 months while on treatment
To collect safety data during the radiation therapy phase | Weekly during radiation therapy
  EKG's will be done once per week and labs twice per week during radiation therapy phase to evaluate safety data.
To evaluate a potential surrogate marker for outcomes | At baseline, before and after radiation therapy, and every 2 cycles during chemotherapy
  Blood will be drawn to analyze methylation patterns as a surrogate marker for outcomes at baseline, before and after radiation therapy, and every 2 cycles during chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Raizer, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Edward Cancer Center, Naperville, Illinois